CLINICAL TRIAL: NCT07361887
Title: Deciphering the Effect of Moderate Wine Consumption on Healthy Aging Through Postprandial Extracellular Vesicles
Acronym: (WINEVOME)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Sergio Montserrat de la Paz, Full Professor, University of Seville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2024-2934
Record Dates: First submitted 2025-12-02; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Atherosclerosis Cardiovascular Disease; Obesity; Metabolic Syndrome; Metabolic Disorders; Inflammation; Neurodegeneration; Neurodegenerative Disease; Alzheimer s Disease
Keywords: blood-brain barrier; microglia; extracellular vesicles; lipidome; proteome; vascular disease
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Metabolic Diseases; Inflammation; Nerve Degeneration; Neurodegenerative Diseases; Vascular Diseases | interventions — Water

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Red Wine (Experimental): Participants will consume red wine (Cabernet Sauvignon) at a dose of 4 mL per kg body weight within 15 minutes. Blood samples will be collected at fasting (0 h), postprandial peak (1-2 h), and post-peak (6 h).
  Interventions: Dietary Supplement: Red Wine
- White Wine (Experimental): Participants will consume white wine (Chardonnay) at a dose of 4 mL per kg body weight within 15 minutes. Blood samples will be collected at fasting (0 h), postprandial peak (1-2 h), and post-peak (6 h).
  Interventions: Dietary Supplement: White Wine
- Water (Control) (Placebo Comparator): Participants will consume water (4 mL per kg body weight) within 15 minutes, serving as the control condition. Blood samples will be collected at fasting (0 h), postprandial peak (1-2 h), and post-peak (6 h).
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: White Wine — Chardonnay, 4 mL/kg body weight
  Arms: White Wine
Dietary Supplement: Red Wine — Cabernet Sauvignon, 4 mL/kg body weight
  Arms: Red Wine
Dietary Supplement: Water — Still water, 4 mL/kg body weight
  Arms: Water (Control)

SUMMARY:
This study aims to investigate how moderate wine consumption influences circulating extracellular vesicles (EVs) in healthy adults. EVs are small particles released by cells that carry proteins, lipids, and genetic material, and play important roles in communication between cells. Participants will consume a single serving of red or white wine, and blood samples will be collected before and after consumption to study changes in the composition and function of EVs. The study will also assess how these EVs affect vascular, immune, and brain-related cells. The results are expected to improve our understanding of how moderate wine intake contributes to cardiovascular and brain health.

DETAILED DESCRIPTION:
Dietary interventions have been consistently proposed as a part of a comprehensive strategy to lower the incidence and severity of atherosclerosis and coronary vascular disease. According to the Dietary Guidelines for Americans 2015-2020, moderate red wine consumption-defined as up to two units of alcohol per day for men and up to one unit of alcohol per day for women-significantly reduces the risk of cardiovascular disease (CVD). Wine is a complex matrix consisting primarily of water (86%) and ethyl alcohol (12%), as well as other different molecules, such as polyphenols, organic acids, tannins, compound minerals, vitamins and biologically active compounds. While most of the nutritional studies have focused on elucidating the mechanisms by which biologically active compounds directly affect cardiovascular-related events, little or nothing is known about the regulatory effect of wine consumption on extracellular vesicles (EVs). EVs are small phospholipid particles that convey molecular bioactive cargoes and play essential roles in intercellular communication and, hence, a multifaceted role in health and disease. Recent advances in research on EVs have significantly enhanced their potential as therapeutic agents for neurological diseases. Owing to their therapeutic properties and ability to cross the blood-brain barrier (BBB), extracellular vesicles are recognized as promising drug delivery vehicles (e.g. polyphenols) for various neurological conditions. For the first time, the purpose of this project is to establish whether the moderate wine consumption may alter the structure, cargo, and functionality of postprandial EVs. In the precision nutrition era, we expect to offer a new insight on EVs and their relationship with wine through the following objectives: 1) To map changes in the lipidome, proteome, polyphenolic cargo, and functional properties of circulating EVs in healthy subjects both at fasting and at postprandial state upon a challenge of a one unit of red or white wine; 2) To analyse the effect of postprandial EVs on atherosclerotic-related events in endothelial and immune cells. 3) To analyse the effect of postprandial EVs on healthy ageing in blood-brain barrier and microglial cells. Collectively, this project will provide fundamental insight into EV biology and remarks the clinical and functional relevance and consequences of moderate wine consumption in health and disease.

ELIGIBILITY:
Inclusion Criteria

* Healthy adult men and women aged 35 to 65 years.
* Body Mass Index (BMI) between 18.5 and 29.9 kg/m².
* Non-smokers or ex-smokers for at least 12 months.
* Moderate alcohol consumers, defined as ≤2 units/day for men and ≤1 unit/day for women.
* Normal fasting glucose and lipid profile at screening.
* Willing and able to refrain from alcohol, polyphenol-rich foods, and intense exercise for 48 hours before each study visit.
* Able to understand the study procedures and provide written informed consent.

Exclusion Criteria

* History or clinical evidence of cardiovascular, hepatic, renal, thyroid, gastrointestinal, or metabolic diseases (including diabetes, dyslipidemia, or hypertension).
* Use of medications or supplements known to affect glucose, lipid, or inflammatory metabolism (e.g., statins, corticosteroids, anti-inflammatory drugs).
* Pregnancy or breastfeeding.
* Recent blood donation (within the last 3 months) or planned blood donation during the study period.
* Major weight change (>5% of body weight) within the last 3 months.
* Participation in another clinical or biomedical study within the previous 3 months.
* Known allergy or intolerance to wine, alcohol, or its components (e.g., sulfites).
* History of alcohol abuse or inability to abstain from alcohol outside the study context.
* Reluctance to receive information about incidental health findings arising from the study.
* Any condition judged by the investigators to limit compliance or increase study risk (e.g., psychiatric disorders, inability to adhere to fasting requirements).

Ages: 35 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of circulating extracellular vesicles | Baseline (0 hours), postprandial peak (2 hours after beverage intake), and post-peak (6 hours after beverage intake).
  Concentration of plasma-derived extracellular vesicles measured after acute intake of red wine, white wine, or water. Extracellular vesicles will be isolated by immunoaffinity methods and quantified using nanoparticle-based analysis. Results will be expressed as particles per milliliter (particles/mL).
Mean size of circulating extracellular vesicles | Baseline (0 hours), postprandial peak (2 hours after beverage intake), and post-peak (6 hours after beverage intake).
  Mean diameter of plasma-derived extracellular vesicles measured after acute intake of red wine, white wine, or water. Extracellular vesicle size will be assessed using dynamic light scattering. Results will be expressed in nanometers (nm).

SECONDARY OUTCOMES:
Postprandial changes in extracellular vesicle proteome | Baseline (0 hours), postprandial peak (2 hours after beverage intake), and post-peak (6 hours after beverage intake).
  Postprandial changes in the protein composition of plasma-derived extracellular vesicles following acute intake of red wine, white wine, or water. EV-associated proteins will be analyzed using quantitative liquid chromatography-tandem mass spectrometry (LC-MS/MS). Results will be expressed as normalized protein abundance.
Postprandial changes in extracellular vesicle lipidome | Baseline (0 hours), postprandial peak (2 hours after beverage intake), and post-peak (6 hours after beverage intake).
  Postprandial changes in the lipid composition of plasma-derived extracellular vesicles following acute intake of red wine, white wine, or water. EV-associated lipid species will be analyzed using quantitative lipidomics by liquid chromatography-mass spectrometry (LC-MS). Results will be expressed as normalized lipid abundance.
Change from baseline in plasma glucose concentration | Baseline (0 hours), 2 hours, and 6 hours after beverage intake
  Venous blood plasma glucose concentration measured using a validated clinical chemistry assay (enzymatic method). Primary metric is change from baseline at each postprandial time point (time point value minus baseline value).
  Unit of Measure: mg/dL
Change from baseline in plasma insulin concentration | Baseline (0 hours), 2 hours, and 6 hours after beverage intake
  Venous blood plasma insulin concentration measured using a validated immunoassay. Primary metric is change from baseline at each postprandial time point (time point value minus baseline value).
  Unit of Measure: µIU/mL
Change from baseline in plasma triglyceride concentration | Baseline (0 hours), 2 hours, and 6 hours after beverage intake
  Venous blood plasma triglyceride concentration measured using a validated clinical chemistry assay (enzymatic method). Primary metric is change from baseline at each postprandial time point (time point value minus baseline value).
  Unit of Measure: mg/dL
Change from baseline in plasma total cholesterol concentration | Baseline (0 hours), 2 hours, and 6 hours after beverage intake
  Venous blood plasma total cholesterol concentration measured using a validated clinical chemistry assay (enzymatic method). Primary metric is change from baseline at each postprandial time point (time point value minus baseline value).
  Unit of Measure: mg/dL
Change from baseline in plasma HDL cholesterol concentration | Baseline (0 hours), 2 hours, and 6 hours after beverage intake
  Venous blood plasma HDL cholesterol concentration measured using a validated clinical chemistry assay (enzymatic method). Primary metric is change from baseline at each postprandial time point (time point value minus baseline value).
  Unit of Measure: mg/dL
Change from baseline in plasma LDL cholesterol concentration | Baseline (0 hours), 2 hours, and 6 hours after beverage intake
  Venous blood plasma LDL cholesterol concentration measured using a validated clinical chemistry assay (enzymatic method). Primary metric is change from baseline at each postprandial time point (time point value minus baseline value).
  Unit of Measure: mg/dL
Change from baseline in plasma interleukin-6 (IL-6) concentration | Baseline (0 hours), 2 hours, and 6 hours after beverage intake
  Venous blood plasma IL-6 concentration measured using a validated immunoassay. Primary metric is change from baseline at each postprandial time point (time point value minus baseline value).
  Unit of Measure: pg/mL
Change from baseline in plasma tumor necrosis factor alpha (TNF-α) concentration | Baseline (0 hours), 2 hours, and 6 hours after beverage intake
  Venous blood plasma TNF-α concentration measured using a validated immunoassay. Primary metric is change from baseline at each postprandial time point (time point value minus baseline value).
  Unit of Measure: pg/mL
Change from baseline in plasma interleukin-1 beta (IL-1β) concentration | Baseline (0 hours), 2 hours, and 6 hours after beverage intake
  Venous blood plasma IL-1β concentration measured using a validated immunoassay. Primary metric is change from baseline at each postprandial time point (time point value minus baseline value).
  Unit of Measure: pg/mL
Change from baseline in plasma monocyte chemoattractant protein-1 (MCP-1/CCL2) concentration | Baseline (0 hours), 2 hours, and 6 hours after beverage intake
  Venous blood plasma MCP-1/CCL2 concentration measured using a validated immunoassay. Primary metric is change from baseline at each postprandial time point (time point value minus baseline value).
  Unit of Measure: pg/mL
Transendothelial electrical resistance (TEER) in an in vitro human blood-brain barrier model after exposure to postprandial extracellular vesicles | EVs isolated at baseline (0 hours) and 2 hours after beverage intake; TEER assessed within 72 hours after EV isolation
  lood-brain barrier (BBB) integrity assessed by transendothelial electrical resistance (TEER) in a human in vitro BBB model after exposure to extracellular vesicles (EVs) isolated from plasma at baseline (0 hours) and postprandial peak (2 hours).
  Unit of Measure: Ω·cm²
Claudin-5 (CLDN5) protein expression in an in vitro human blood-brain barrier model after exposure to postprandial extracellular vesicles | EVs isolated at baseline (0 hours) and 2 hours after beverage intake; protein expression assessed within 72 hours after EV isolation
  Tight junction protein expression assessed in the BBB model by Claudin-5 (CLDN5) protein abundance after exposure to EVs isolated at baseline (0 hours) and 2 hours post intake. Protein expression quantified using immunoblotting or immunofluorescence and reported relative to the control condition.
  Unit of Measure: Fold change (dimensionless)
Occludin (OCLN) protein expression in an in vitro human blood-brain barrier model after exposure to postprandial extracellular vesicles | EVs isolated at baseline (0 hours) and 2 hours after beverage intake; protein expression assessed within 72 hours after EV isolation
  Tight junction protein expression assessed in the BBB model by occludin (OCLN) protein abundance after exposure to EVs isolated at baseline (0 hours) and 2 hours post intake. Protein expression quantified using immunoblotting or immunofluorescence and reported relative to the control condition.
  Unit of Measure: Fold change (dimensionless)
Interleukin-6 (IL-6) concentration in microglial culture supernatant after exposure to postprandial extracellular vesicles | EVs isolated at baseline (0 hours) and 2 hours after beverage intake; cytokines assessed within 72 hours after EV isolation
  Microglial activation assessed by IL-6 concentration in culture supernatant after exposure to EVs isolated at baseline (0 hours) and 2 hours post intake. Cytokine concentration quantified using a validated immunoassay.
  Unit of Measure: pg/mL
Tumor necrosis factor alpha (TNF-α) concentration in microglial culture supernatant after exposure to postprandial extracellular vesicles | EVs isolated at baseline (0 hours) and 2 hours after beverage intake; cytokines assessed within 72 hours after EV isolation
  Microglial activation assessed by TNF-α concentration in culture supernatant after exposure to EVs isolated at baseline (0 hours) and 2 hours post intake. Cytokine concentration quantified using a validated immunoassay.
  Unit of Measure: pg/mL
IL1B mRNA expression in microglia after exposure to postprandial extracellular vesicles | EVs isolated at baseline (0 hours) and 2 hours after beverage intake; gene expression assessed within 72 hours after EV isolation
  Microglial activation assessed by IL1B mRNA expression after exposure to EVs isolated at baseline (0 hours) and 2 hours post intake. Gene expression quantified by RT-qPCR and reported as relative expression versus control condition.
  Unit of Measure: Fold change (dimensionless)
Endothelial VCAM-1 protein expression after exposure to postprandial extracellular vesicles | EVs isolated at baseline (0 hours) and 2 hours after beverage intake; assays conducted within 48 hours after EV isolation
  Endothelial activation assessed by VCAM-1 protein expression in cultured human umbilical vein endothelial cells after exposure to extracellular vesicles isolated from plasma at baseline (0 hours) and postprandial peak (2 hours). Protein expression quantified by immunoblotting or immunofluorescence and reported relative to control condition.
  Unit of Measure: Fold change (dimensionless)
Polyphenolic content of extracellular vesicles after wine intake | Baseline (0 hours), postprandial peak (2 hours after beverage intake), and post-peak (6 hours after beverage intake).
  Identification and quantification of polyphenolic compounds encapsulated within plasma-derived extracellular vesicles following acute intake of red wine or white wine. Polyphenols will be analyzed using ultra-high-performance liquid chromatography coupled to quadrupole-Orbitrap mass spectrometry. Results will be expressed as normalized peak areas and concentrations relative to internal standards.
Spearman correlation between EV cargo score and change from baseline in plasma glucose concentration | Baseline (0 hours), 2 hours, and 6 hours after beverage intake (plasma glucose); EVs isolated at baseline (0 hours) and 2 hours after beverage intake
  Association assessed using Spearman rank correlation (ρ) between EV cargo score (PC1 derived from normalized EV proteomic and lipidomic features measured by mass spectrometry) and the systemic response measure defined as change from baseline in plasma glucose concentration at postprandial time points. The outcome measure is Spearman's ρ.
  Unit of Measure: Spearman's ρ (dimensionless)
Endothelial ICAM-1 protein expression after exposure to postprandial extracellular vesicles | EVs isolated at baseline (0 hours) and 2 hours after beverage intake; assays conducted within 48 hours after EV isolation
  Endothelial activation assessed by ICAM-1 protein expression in cultured human umbilical vein endothelial cells after exposure to extracellular vesicles isolated from plasma at baseline (0 hours) and postprandial peak (2 hours). Protein expression quantified by immunoblotting or immunofluorescence and reported relative to control condition.
  Unit of Measure: Fold change (dimensionless)
Nitric oxide (NO) production in endothelial cell culture supernatant after exposure to postprandial extracellular vesicles | EVs isolated at baseline (0 hours) and 2 hours after beverage intake; assays conducted within 48 hours after EV isolation
  Endothelial response assessed by nitric oxide production after exposure to extracellular vesicles isolated from plasma at baseline (0 hours) and postprandial peak (2 hours). NO production quantified in culture supernatant using a validated colorimetric assay (e.g., nitrite/nitrate).
  Unit of Measure: µM

CONTACTS AND LOCATIONS:
Locations (1):
- Av. de Sánchez Pizjuán, s/n, 41009 Sevilla Facultad de Medicina . Universidad de Sevilla, Seville, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: Undecided